CLINICAL TRIAL: NCT05968365
Title: Clinical Trial of the Safety and Effectiveness of Vision Pro Electronic Blind Aid Device
Brief Title: Evaluate the Safety and Effectiveness of Electronic Vision-aid Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wicab Technologies (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WKKJ-2020001
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2021-12

CONDITIONS: the Blind

STUDY DESIGN:
Intervention Model Description: The clinical trial was a prospective, single-group, uncontrolled design using the target value method
  Three centers participated
  A total of 36 patients were enrolled. It was developed and produced by Weikan Technology in subjects who agreed to be enrolled
  The "Vision Pro" is trained, and after no less than 3 hours of training, the subject is good at it
  Evaluate the safety and effectiveness of obstacle perception and recognition in the process of walking, and evaluate the test product in auxiliary sight
  Safety and effectiveness of obstacle perception and recognition for disabled walkers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: electronic Vision-aid Device — Electronic blind aid is a non-invasive electronic aid product for the visually impaired. The product converts visual signals into tactile signals. The Vision Pro is designed for people with poor or no visual perception. The product does not change the previous travel mode of the visually impaired, and provides additional external information for the visually impaired on the basis of their existing cognition. The product can provide the visually impaired person with additional external information based on the cognition in front of them. The product can feedback the environmental information within 2.52.5 meters in front of the visually impaired person in the form of electrical stimulation to the visually impaired person. The visually impaired person can be stimulated by the tongue current to help them identify obstacles and give early warning. Avoid obstacles and give early warning.

SUMMARY:
To evaluate the safety and effectiveness of electronic Vision-aid Device in walking and obstacle recognition for visually blind people

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 (including 18 and 65 years old)；
2. Visually impaired people；
3. Primary blind and visually impaired people
4. visual acuity is no light ~ < 0.02；
5. visual field radius less than 5°);

Exclusion Criteria:

1. . Allergic to nickel or stainless steel;
2. epileptic seizures;
3. pregnant women； 4.、implanted with electronic medical devices ；

5、 intellectual disability ； 6、 mental illness; 7、 Oral diseases； 8、oral ulcers, herpes, herpes simplex, oral thrush and map tongue； 9、 speech dysfunction, 10、limited mobility and hearing impairment;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
obstacle identification | 40 minutes
  The success rate of obstacle identification

SECONDARY OUTCOMES:
obstacle avoidance test | 40 minutes
  the success rate of obstacle avoidance

CONTACTS AND LOCATIONS:
Locations (1):
- Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
ResMan